CLINICAL TRIAL: NCT07238244
Title: Development and Validation of a Machine Learning-Based Risk Prediction Model for Recurrence After Percutaneous Balloon Compression in Trigeminal Neuralgia Patients: A Retrospective Cohort Study
Brief Title: Risk Factors for Recurrence of Trigeminal Neuralgia After Percutaneous Balloon Compression
Status: Not yet recruiting | Type: Observational
Sponsor: Second Xiangya Hospital of Central South University (Other)
Collaborators: Yueyang Hospital of Traditional Chinese Medicine (Unknown)
Responsible Party: Principal Investigator, YaPing Wang, Professor, Second Xiangya Hospital of Central South University
Other Study IDs: LYF2022139
Record Dates: First submitted 2025-09-30; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-09

CONDITIONS: Trigeminal Neuralgia
Keywords: Trigeminal Neuralgia; Percutaneous Balloon Compression; predication; Machine Learning Model
MeSH Terms: conditions — Trigeminal Neuralgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Percutaneous Balloon Compression — The intervention studied is Percutaneous Balloon Compression (PBC). It is a minimally invasive surgical intervention used for the treatment of primary trigeminal neuralgia (TN), which involves percutaneously inserting a balloon to compress the trigeminal ganglion, aiming to relieve pain in patients with TN who are unresponsive to drug therapy or unable to tolerate drug adverse reactions.

SUMMARY:
The goal of this observational study is to develop and validate a machine learning-based model for predicting pain recurrence risk after percutaneous balloon compression (PBC) in adult patients with primary trigeminal neuralgia (TN) who had their first PBC treatment. The main questions it aims to answer are:

Can the machine learning-based model accurately predict pain recurrence after PBC in these primary TN patients? What key factors (like patient baseline traits, imaging parameters, surgical operation data) affect PBC post-operative pain recurrence? Do machine learning algorithms perform better than traditional Cox proportional hazards regression in predicting such recurrence? Participants (with existing PBC treatment records) will have their past data-including clinical info from the hospital's electronic medical record system, imaging data from the image archiving system, surgical data from the surgical anesthesia system, and follow-up data from the outpatient system-collected and analyzed to build and validate the prediction model.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 18 years.
2. Meet the diagnostic criteria for primary trigeminal neuralgia according to the International Classification of Headache Disorders, 3rd edition (ICHD-3).
3. Undergo the first PBC treatment.
4. Have complete preoperative clinical data, imaging data, and intraoperative records.
5. Have at least one postoperative follow-up record available for determining the recurrence status.

Exclusion Criteria:

1. Secondary trigeminal neuralgia (e.g., caused by cerebellopontine angle tumors, multiple sclerosis, etc.).
2. Missing rate of key predictor variables (e.g., balloon shape) or outcome variables > 15%.
3. Postoperative loss to follow-up (defined as no follow-up records available).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (aged ≥ 18 years) who underwent percutaneous balloon compression (PBC) with primary trigeminal neuralgia (TN) who had their first PBC treatment at the Department of Pain Medicine, the Second Xiangya Hospital of Central South University between January 2018 and June 2025, and were willing to participate in postoperative follow-up were selected as the study subjects
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Pain Recurrence After Percutaneous Balloon Compression in Patients with Primary Trigeminal Neuralgia | through study completion, an average of 3 year
  The primary outcome measure focuses on whether pain recurrence occurs in patients with primary TN after their first PBC treatment, defined as a dichotomous variable ("recurred" or "not recurred").
  Recurrence Criteria: Postoperative pain intensity, as assessed by the Barrow Neurological Institute Pain Intensity Score, rebounds to Grade IV ("persistent pain controllable with medication") or Grade V ("severe pain uncontrollable with medication"), and this pain status persists for at least 1 week. Additionally, the recurrence must be accompanied by the need to increase the dose of pain medication or undergo reinterventional treatment (e.g., repeated PBC or other surgical procedures) to manage the pain.

IPD SHARING:
Plan to Share IPD: Yes
The Individual Participant Data (IPD) to be shared in this study will be strictly de-identified (with all personal identifiers such as names, ID numbers, hospital admission numbers, and contact information removed and replaced with unique study serial numbers) and limited to data relevant to verifying the research objectives.Raw imaging files, full electronic medical records, and any sensitive data unrelated to the study's prediction model verification will not be included in the shared IPD to ensure participant privacy and data security.
Supporting Information: Study Protocol, SAP

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-07-30): https://cdn.clinicaltrials.gov/large-docs/44/NCT07238244/Prot_SAP_000.pdf